CLINICAL TRIAL: NCT01889316
Title: Performance Comparison of a New Fetal/Maternal Monitor With an FDA-cleared Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Meg Hill, Principal Investigator, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-0197; FWA00004218 (Other: Monica Healthcare); NCT02041949 (obsolete NCT alias)
Record Dates: First submitted 2013-05-01; First posted 2013-06-28 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Labor Fetal Anoxia
Keywords: Fetal monitoring; ECG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AN24 in addition to new device (Novii) (Other): FDA-cleared device (The AN24 device) used in conjunction with the new device (Novii).
  Both devices will be placed on the patient's abdomen. Hence the patient acts as their own control.
  Interventions: Device: Novii; Device: AN24

INTERVENTIONS:
Device: Novii — The Novii is a modified device with similar technology to the AN24 device already being used in the USA.
Device: AN24

SUMMARY:
This is a prospective clinical trial involving the use of the FDA-cleared Fetal ECG tracing in labor with the AN24 (Fetal Monitoring device marketed by Monica Healthcare) to the Novii (a newer device also created by Monica Healthcare) using the same technology with different monitor placement.

DETAILED DESCRIPTION:
This study has one arm, in which Both the FDA - Approved AN24 (Fetal Monitoring device marketed by Monica Healthcare) and the new device (Novii, being investigated in this clinical trial) will be placed on the patient's abdomen. After delivery of the patient's infant, the data will be abstracted from the second device. This data will be compared to the data from the first device for accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Term Laboring Patients

Exclusion Criteria:

* Preterm Labor
* Fetal Anomaly
* Imminent cesarean

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of the Novii when compared to the AN24 | duration of the patient's labor
  Both the AN24 device and the Novii device will be placed on the patient's abdomen at the same time. After the patient has delivered their infant, the data from the Novii will be downloaded and checked against that from the AN24 to assess for accuracy of fetal monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Meg Hill, MBBS, Principal Investigator — University of Arizona
Locations (1):
- University Medical Center, Tucson, Arizona, United States